CLINICAL TRIAL: NCT06693115
Title: The Use of Continuous Glucose Monitoring With Patients Undergoing a New Subcutaneous Insulin Protocol for Mild to Moderate Diabetic Ketoacidosis or Hyperosmolar Hyperglycemic State
Brief Title: Continuous Glucose Monitoring Using a New Subcutaneous Insulin Protocol for Mild to Moderate Diabetic Ketoacidosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A24-338
Record Dates: First submitted 2024-11-06; First posted 2024-11-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Ketoacidosis; Hyperglycemia
MeSH Terms: conditions — Diabetic Ketoacidosis; Hyperglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CGM with alerts (Experimental): The experimental group will have a Dexcom 7 CGM placed by a trained and credentialed member of the research team, or by a trained care team member (e.g. nurse, physician, diabetes educator).
  CGM devices will be set to alert the care team when interstitial glucose levels hit 250 mg/dL and 150 mg/dL. Dexcom 7s automatically alert when glucose levels are 55 mg/dL or lower. Nurses will be instructed to check the glucose trends on the CGM device when alerted. They will be asked to check glucose levels with a FSBG according to the following instructions:
  1. CGM alerts to interstitial glucose level of 250 mg/dL AND trend indicates rapidly decreasing glucose levels
  2. CGM alerts to interstitial glucose level of 150 mg/dL or less.
  Interventions: Device: CGM with alerts
- CGM without alerts (No Intervention): The control group will have a Dexcom 7 CGM placed by a trained and credentialed member of the research team, or by a trained care team member (e.g. nurse, physician, diabetes educator).
  The control group will have the device placed and glucose levels will be collected, but the device will not be set to alert (though note that the Dexcom 7 CGM will always alert when glucose drops below 55 mg/dl, so this alert will exist for both groups).

INTERVENTIONS:
Device: CGM with alerts — CGM devices will be set to alert the care team when interstitial glucose levels hit 250 mg/dL and 150 mg/dL. Dexcom 7s automatically alert when glucose levels are 55 mg/dL or lower. Nurses will be instructed to check the glucose trends on the CGM device when alerted. They will be asked to check glucose levels with a FSBG according to the following instructions:
  1. CGM alerts to interstitial glucose level of 250 mg/dL AND trend indicates rapidly decreasing glucose levels (indicated by double down arrow on Dexcom 7)
  2. CGM alerts to interstitial glucose level of 150 mg/dL or less.
  Arms: CGM with alerts

SUMMARY:
Using a prospective, mixed methods study design, the investigators will assess the feasibility, usefulness, and care team acceptability of CGM in conjunction with FSBG during implementation of the new subQ DKA/HHS protocol at Regions Hospital. This will include evaluating how many patients agree to have a CGM device placed, time to place the CGM devices, CGM impact on length of stay, level of care required, frequency of alerts to changing glucose levels events, and assessing the match between CGM and FSBG readings done in the inpatient setting. Results will help inform cost effective, safe, patient-centered strategies, while gauging care team satisfaction to optimize DKA and HHS management in the future.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) and Hyperosmolar Hyperglycemic State (HHS) are severe complications of diabetes mellitus and one of the most common causes of hospital admission among people with diabetes. Up to now, the standard of care for managing DKA and HHS at Regions Hospital has involved intravenous (IV) insulin to treat hyperglycemia. However, the use of IV insulin is associated with increased care team resource utilization and the potential for adverse events such as hypoglycemia. Regions Hospital is in the process of implementing a new subcutaneous (subQ) insulin protocol, which has the potential to reduce resource utilization and improve patient safety, while producing similar outcomes for patients. One critical part of the new protocol is reducing the frequency of point of care capillary blood glucose monitoring, commonly known as a Finger Stick Blood Glucose test (FSBG) from hourly (Q1) to every 4 hours (Q4). The use of subQ insulin with less frequent blood sugar monitoring is possible owing to subQ insulin's slower mechanism of action than the IV insulin. Protocols have been shown to be safe within other hospital systems. However, the change from Q1 to Q4 monitoring of blood sugars does lead to some concern on the part of providers about correcting hyperglycemia too slowly or failing to recognize impending hypoglycemic events.

The use of Continuous Glucose Monitoring (CGM) technology has been proposed to provide continuous (i.e. every 5 mins) updates about patient glucose levels in between FSBG checks in patients being treated for mild to moderate DKA or HHS. This continuous monitoring would help provide prompt identification of hypoglycemic episodes and improve safety during hospitalization, a change that could provide peace of mind to care providers and patients as the change is made from Q1 to Q4 FSBG.

Using a prospective, mixed methods study design, the investigators will assess the feasibility, usefulness, and care team acceptability of CGM in conjunction with FSBG during implementation of the new subQ DKA/HHS protocol at Regions Hospital. This will include evaluating how many patients agree to have a CGM device placed, time to place the CGM devices, CGM impact on length of stay, level of care required, frequency of alerts to changing glucose levels events, and assessing the match between CGM and FSBG readings done in the inpatient setting. Results will help inform cost effective, safe, patient-centered strategies, while gauging care team satisfaction to optimize DKA and HHS management in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presents at Regions Hospital ED including transfers from other hospitals
* Meets criteria for new subQ insulin protocol:
* Diagnosis of DKA or HHS (hyperosmolar hyperglycemic state) and provider decision to initiate insulin
* pH ≥ 7.1
* HCO3 ≥ 12

Exclusion Criteria:

* Under 18 years of age
* Excluded from new subQ protocol, specifically:
* Acute CHF exacerbation
* Acute MI (ACS/NSTEMI type 1 not demand ischemia)
* CKD stage 4 or AKI with creatinine > 3
* ESLD
* Pregnancy
* Severe sepsis or septic shock
* AMS > if patient cannot consent
* Euglycemic DKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility of CGM placement by hospital staff for patients experiencing hyperglycemia | Duration of hospital stay from admission to discharge (average of 4 days).
  Recruitment, overall participation, and completion rate.
Determine feasibility of CGM placement by hospital staff for patients experiencing hyperglycemia | From time of admission until the time of first insulin administration by CGM (average of 2 hours).
  Time to place CGM (time from admission, time from insulin administration).

SECONDARY OUTCOMES:
Evaluate patient safety and care outcomes related to use of CGM during hospitalization | Duration of hospital stay from admission to discharge (average of 4 days).
  Length of hospital stay (ED, ICU, and/or Non-ICU)
Evaluate patient safety and care outcomes related to use of CGM during hospitalization | From admission to medical clearance for discharge or transfer to another healthcare facility, whichever comes first (average of 4 days).
  Time until DKA/HHS resolution
Describe accuracy and usefulness of CGM for monitoring resolution from hyperglycemia | Duration of hospital stay from admission to discharge (average of 4 days).
  Hits: how often does CGM device alert to glucose levels that are confirmed by FSBG to require intervention?
  Misses: how often does FSBG identify glucose levels that require intervention when CGM does not alert?
  False alarms: how often does CGM device alert when FSBG suggests no intervention is necessary?
  Nurse acceptability of CGM use:
  The investigators seek to measure care team acceptability of CGM during the treatment of patients with DKA/HHS by comparing their survey responses in reference to caring for patients who have CGM devices with alerts (Experimental group) vs patients who have CGM devices without alerts (Control group).

CONTACTS AND LOCATIONS:
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to for HIPAA considerations and data is only to be used for measurement of site-specific protocols.

REFERENCES:
- [Background] Wallia A, Umpierrez GE, Nasraway SA, Klonoff DC; PRIDE Investigators. Round Table Discussion on Inpatient Use of Continuous Glucose Monitoring at the International Hospital Diabetes Meeting. J Diabetes Sci Technol. 2016 Aug 22;10(5):1174-81. doi: 10.1177/1932296816656380. Print 2016 Sep. PMID 27286715
- [Background] Park E, Kim M. Clinical Use of Continuous Glucose Monitoring in Critically Ill Pediatric Patients with Diabetic Ketoacidosis. Diabetes Technol Ther. 2023 Aug;25(8):529-537. doi: 10.1089/dia.2023.0012. Epub 2023 Jul 17. PMID 37155338
- [Background] Klonoff DC, Ahn D, Drincic A. Continuous glucose monitoring: A review of the technology and clinical use. Diabetes Res Clin Pract. 2017 Nov;133:178-192. doi: 10.1016/j.diabres.2017.08.005. Epub 2017 Sep 1. PMID 28965029
- [Background] Faulds ER, Jones L, McNett M, Smetana KS, May CC, Sumner L, Buschur E, Exline M, Ringel MD, Dungan K. Facilitators and Barriers to Nursing Implementation of Continuous Glucose Monitoring (CGM) in Critically Ill Patients With COVID-19. Endocr Pract. 2021 Apr;27(4):354-361. doi: 10.1016/j.eprac.2021.01.011. Epub 2021 Jan 27. PMID 33515756
- [Background] Zelada H, Perez-Guzman MC, Chernavvsky DR, Galindo RJ. Continuous glucose monitoring for inpatient diabetes management: an update on current evidence and practice. Endocr Connect. 2023 Sep 25;12(10):e230180. doi: 10.1530/EC-23-0180. Print 2023 Oct 1. PMID 37578799
- [Background] Wright JJ, Williams AJ, Friedman SB, Weaver RG, Williams JM, Hodge E, Fowler M, Bao S. Accuracy of Continuous Glucose Monitors for Inpatient Diabetes Management. J Diabetes Sci Technol. 2023 Sep;17(5):1252-1255. doi: 10.1177/19322968221076562. Epub 2022 Feb 7. PMID 35128974